CLINICAL TRIAL: NCT00308087
Title: Randomized, Open Label, Phase II Trial Comparing Rituximab Plus Sargramostim to Rituximab Monotherapy for the Treatment of Relapsed Follicular B-cell Lymphoma
Brief Title: Comparison Study of Rituximab Plus Sargramostim to Rituximab Alone for Relapsed Follicular B-cell Lymphoma, a Form of Non-Hodgkin's Lymphoma
Acronym: PREMIER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated by sponsor due to low enrollment; see details below
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 310421; 91499 (Other: Genzyme); PREMIER (Other: Genzyme)
Record Dates: First submitted 2006-03-28; First posted 2006-03-29 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma, Follicular
Keywords: Sargramostim; Leukine; NHL
MeSH Terms: conditions — Lymphoma, Follicular | interventions — sargramostim; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Active Comparator)
  Interventions: Drug: Rituximab
- Rituximab + Sargramostim (Experimental)
  Interventions: Drug: Sargramostim (Leukine); Drug: Rituximab

INTERVENTIONS:
Drug: Sargramostim (Leukine) — Sargramostim 250 μg, administered subcutaneously (SC) 3 times weekly for 8 weeks, beginning at least 1 hour before the first dose of rituximab
  Other Names: Sargramostim; Leukine; Bay86-5326
  Arms: Rituximab + Sargramostim
Drug: Rituximab — Four doses of rituximab 375 mg/m2, administered intravenously (IV) once weekly for 4 weeks

SUMMARY:
The purpose of this study is to evaluate whether treatment with rituximab plus sargramostim will be more effective than rituximab alone.

DETAILED DESCRIPTION:
On 29 May 2009, Bayer began transitioning the sponsorship of this trial to Genzyme. As of 29 August 2009, Genzyme assumed responsibility for the close out of the study. NOTE: This study was originally posted by sponsor Berlex, Inc. Berlex, Inc. was renamed to Bayer HealthCare, Inc.

The study was terminated early due to low enrollment; significant changes to the protocol would have been required to keep pace with the changing therapeutic landscape of indolent lymphoma.

ELIGIBILITY:
Inclusion Criteria (abbreviated list):

* Relapsed follicular B-cell lymphoma
* One or more previous therapies for non-Hodgkin's
* At least one measurable tumor by CT scan or MRI
* Additional criteria to be determined at screening visit

Exclusion Criteria (abbreviated list):

* Rituximab refractory (less than 6 months from last treatment with rituximab to relapse)
* Currently receiving treatment for another cancer
* Infection currently being treated
* Active Hepatitis B
* History of HIV infection
* Pregnant
* Additional criteria to be determined at screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (22):
- United States (21):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Los Angeles, California
  - Montebello, California
  - Pleasant Hill, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Elk Grove Village, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - New Albany, Indiana
  - Duluth, Minnesota
  - Fresh Meadows, New York
  - New York, New York
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Houston, Texas
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred ninety-six (196) patients were planned and 44 centers were open for enrollment. Eighty-two (82) patients were screened from 22 investigator sites across the United States and Puerto Rico.
Pre-assignment Details: 82 patients screened
Groups:
- Rituximab + Sargramostim: Sargramostim 250 μg, administered subcutaneously (SC) 3 times weekly for 8 weeks, beginning at least 1 hour before the first dose of rituximab. Plus four doses of rituximab 375 mg/m2, administered intravenously (IV) once weekly for 4 weeks.
Period: Overall Study
Arm/Group | Rituximab | Rituximab + Sargramostim
Started | 37 | 38
Completed | 1 (Completers finished treatment and the 24 month follow-up.) | 1 (Completers finished treatment and the 24 month follow-up.)
Not Completed | 36 | 37
Not completed — Progressive Disease | 19 | 21
Not completed — Study Closure | 11 | 12
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Rituximab + Sargramostim | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.23) | 59.4 (8.68) | 60.5 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 16 | 20 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 26 | 29 | 55
  Black | 2 | 4 | 6
  Hispanic | 7 | 3 | 10
  Asian | 1 | 2 | 3
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response or Unconfirmed Complete Response at Week 8 With Confirmation at Week 12
Description: Count of number of participants who responded with a Complete Response (complete disappearance of all detectable clinical and radiological evidence of disease) at week 8 and again clinically and radiologically confirmed at week 12.
Time Frame: Week 8 (confirmed at Week 12)
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 37 | 38
participants | 1 | 3
Statistical Analysis 1: Comparison: Rituximab vs Rituximab + Sargramostim; Test type: Superiority or Other; p = 0.6182, 2-sided Exact Conditional Test — Exact Conditional Test is stratified on the number > of prior therapies (1 or 2, 3 or more prior therapies)

2. Secondary Outcome: Summary of Treatment-Emergent Adverse Events (TEAE)
Description: Count of the number of participants who experienced treatment emergent adverse events (TEAEs). TEAEs occurred during the time study intervention was being taken occurring on or after Day 1 and no longer than 30 days after the last dose of study medication.
Time Frame: up to 12 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 37 | 38
participants
  Patients with TEAEs | 34 | 38
  Patients with Treatment-Related TEAEs | 21 | 37
  Number of Deaths | 0 | 0
  Patients with Serious TEAEs | 4 | 4
  Patients with Study Discontinuation due to TEAEs | 0 | 2

3. Secondary Outcome: Participant Summary of Best Response Across All Visits
Description: Count of participants' best response within categories defined by the International Working Group (IWG):
  > Complete Response (complete disappearance of detectable clinical and radiological evidence of disease),
  > Complete Response Unconfirmed (unconfirmed complete disappearance),
  > Partial Response (>=50% decrease sum of the product of the greatest diameters in the six largest dominant nodes or nodal masses),
  > Stable Disease (neither response nor disease progression),
  > Progression (new lesion or increase by 50% of previously involved sites from nadir).
Time Frame: up to 24 months
Population: Intent to treat population
Measure: Number; unit: participants
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 37 | 38
participants
  Complete Response | 5 | 5
  Complete Response Unconfirmed | 0 | 0
  Partial Response | 13 | 14
  Stable Disease | 11 | 15
  Progression | 4 | 3
  Unknown | 0 | 0

4. Secondary Outcome: Kaplan-Meier Estimates of Progression-Free Survival
Description: Time to event was measured from the date of randomization to the date of first progressive disease (PD) or death.
Time Frame: 24 months
Population: Intent to treat population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 37 | 38
Days | 361.0 [170.0 to 540.0] | 455.0 [238.0 to 549.0]
Statistical Analysis 1: Comparison: Rituximab vs Rituximab + Sargramostim; Log rank analysis is a comparison between treatment groups of the distribution of time to first progressive disease or death; Test type: Superiority or Other; p = 0.5501, Log Rank

5. Secondary Outcome: Kaplan-Meier Estimates for Duration of Partial Response or Better to Treatment
Description: Count of days in which a participant experiences a Partial Response (>=50% decrease sum of the product of the greatest diameters in the six largest dominant nodes or nodal masses) or better. Time to event was measured from the date of response to the date of progressive disease (PD) or death.
Time Frame: 24 months
Population: Intent to treat population.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 18 | 19
Days | 297.0 [264.0 to 642.0] | 396.0 [300.0 to 484.0]
Statistical Analysis 1: Comparison: Rituximab vs Rituximab + Sargramostim; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8217, Log Rank

6. Secondary Outcome: Summary of Cost Effectiveness
Description: A cost-effectiveness analysis from the payer perspective was to be performed. Only direct medical costs for each patient during the study period were to be included for analysis. Costs were to be calculated by multiplying each health care resource unit by the amount reimbursed by a payer. Health care resource utilization units are a way to normalize the quantity of health care provided to each participant so that costs can be compared.
Time Frame: 24 months
Population: No participants were analyzed because the study was terminated early due to low enrollment.
Arm/Group | Rituximab | Rituximab + Sargramostim
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Rituximab | Rituximab + Sargramostim
Serious Adverse Events (participants affected / at risk) | 5/37 | 7/38
Other Adverse Events (participants affected / at risk) | 33/37 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=37) | Rituximab + Sargramostim (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Facial pain (General disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=37) | Rituximab + Sargramostim (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 2
Dry eye (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 14
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oedema mouth (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 2
Chills (General disorders) | 6 | 16
Fatigue (General disorders) | 9 | 12
Feeling abnormal (General disorders) | 1 | 0
Induration (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 1
Infusion related reaction (General disorders) | 3 | 1
Infusion site erythema (General disorders) | 1 | 0
Injection site discolouration (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 9
Injection site haematoma (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 6
Injection site pruritus (General disorders) | 0 | 8
Injection site rash (General disorders) | 0 | 2
Injection site reaction (General disorders) | 0 | 7
Injection site swelling (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 6
Pain (General disorders) | 2 | 5
Pyrexia (General disorders) | 1 | 9
Cytokine release syndrome (Immune system disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 3
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood albumin increased (Investigations) | 0 | 1
Blood immunoglobulin g decreased (Investigations) | 0 | 1
Blood immunoglobulin m decreased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2
White blood cell count increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 7
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 8 | 9
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Tension headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 5
Dysuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3
Flushing (Vascular disorders) | 0 | 2
Hot flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 4
Pallor (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
One hundred ninety-six patients were planned and 75 enrolled prior to termination. The study was terminated early due to low enrollment, and the extent of changes needed to the protocol to keep pace with therapeutic changes for indolent lymphoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to provide sponsor with an advance copy of any proposed publication or presentation at least 60 days prior to the planned submission or presentation. Genzyme shall have 30 days in which to recommend changes and to inform investigator if confidential information is contained. In the event of the latter, investigator will delay or prevent publication for no more that 90 days to permit sponsor to file a patent application.